CLINICAL TRIAL: NCT01016626
Title: Open Label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetic Characteristics of CKD-4101 Tablet, in Healthy Volunteers
Brief Title: Study to Evaluate the Pharmacokinetic Characteristics of CKD-4101 (Mycophenolate Mofetil) Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Ji Hye Lee, Chong Kun Dang Pharmaceutical
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CKD-123HPS08E; 123HPS08E
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Healthy volunteers; Mycophenolate Mofetil
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-4101 tablet (Experimental)
  Interventions: Drug: CKD-4101 tablet
- Mycophenolate Mofetil capsule (Active Comparator)
  Interventions: Drug: Mycophenolate Mofetil capsule

INTERVENTIONS:
Drug: CKD-4101 tablet — CKD-4101 tablet 1000 mg
  * 500mg/tablet, PO, 2 tablet once daily for D1 and D8(crossover)
  Arms: CKD-4101 tablet
Drug: Mycophenolate Mofetil capsule — Mycophenolate Mofetil capsule 1000 mg
  * 250mg/capsule, PO, 4 capsule once daily for D1 and D8(crossover)
  Arms: Mycophenolate Mofetil capsule

SUMMARY:
The purpose of this study is to evaluate safety and tolerance by comparing pharmacokinetic characteristics between the CKD-4101 tablet and Mycophenolate mofetil capsule when administered alone to healthy volunteers.

DETAILED DESCRIPTION:
Healthy volunteers are administrated single-dose over the period I and II (Crossover) of CKD-4101 1000mg and Mycophenolate mofetil capsule 1000mg.

Every time before and after each medication, PK parameters and safety of CKD-4101 tablet and Mycophenolate mofetil capsule is performed using a blood sample and conducting some tests respectively.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 45 aged in healthy males
* Weight more than 45 kg, IBW ± 20% within the range

  * Ideal body weight = (Height cm - 100) x 0.9
* Agreement with written informed consent

Exclusion Criteria:

* Subject has symptoms of acute disease within 28 days of starting administration of investigational drug
* Subject with known for history(such as inflammatory gastrointestinal disease, gastric or duodenal ulcer, liver diseases and so on) which affect the ADME of drug
* Clinically significant, active gastrointestinal system, cardiovascular system, pulmonary system, renal system, Blood system, digestive system, central nervous system, mental disease or malignancy disease.
* Inadequate subject by medical examination(medical history, physical examination,ECG, laboratory test) within 28 days of starting administration of investigational drug
* Inadequate result of laboratory test

  * AST or ALT > 1.25 x upper limit of normal range
  * Total bilirubin > 1.25 x upper limit of normal range
  * Abnormal level of WBC, Platelet, Hemoglobin WBC < 3.5 x 1000/µL PLT < 100 x 1000/µL Hemoglobin < 11g/dL
* Clinically significant allergic disease(Except for mild allergic rhinitis seems to be not need for medication)
* HGPRT(Hypoxanthine-guanine phosphoribosyl-transferase)deficiency patient such as Lesch-Nyhan syndrome and kelley-Seegmiller syndrome
* Severe renal dysfunction: Creatinine clearance less than 50ml/min by cockroft-Gault calculation
* Subject with known for hypersensitivity reaction to mycophenolic acid and mycophenolate mofetil analog
* Previously participated in other trial within 60 days
* Treatment with dug-medicated induction/inhibition metabolic enzyme such as barbiturates within 1month or with may affect the clinical trial within 10 days
* Unusual diet may affect the ADME of drug
* Not able to taking the institutional standard meal
* Previously make whole blood donation within 60 days or component blood donation within 20 days
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking(alcohol > 30 g/day) and during clinical trials can not be drunk or severe heavy smoker (cigarette > 1/2 pack per day)
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of CKD-4101 tablet and Mycophenolate Mofetil capsule. | 0-48 hrs

SECONDARY OUTCOMES:
To evaluate the safety of CKD-4101 tablet and Mycophenolate Mofetil capsule from vital signs, physical exam, ECG, laboratory test, adverse event and so on. | 0-48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, Principal Investigator — jypark21@korea.ac.kr
Locations (1):
- The Korea University Anam Hospital, Seoul, South Korea